CLINICAL TRIAL: NCT01559701
Title: A Long-Term, Open-Label, Safety Study Of PTI-821 In Patients With Moderate To Severe Chronic Low Back Pain Or With Moderate To Severe Chronic Pain Due To Osteoarthritis Of The Hip Or Knee
Brief Title: Long-term Safety of PF-00345439 (Oxycodone)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-821-CM; B4501007
Record Dates: First submitted 2012-03-13; First posted 2012-03-21 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: Pain
Keywords: Safety; PF-00345439; Remoxy; PTI-821
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-00345439 (oxycodone) (Experimental): PF-00345439 (oxycodone)
  Interventions: Drug: PF-00345439

INTERVENTIONS:
Drug: PF-00345439 — 5-80 mg twice-a-day for 12 months
  Other Names: PTI-821, Remoxy

SUMMARY:
Long-Term Safety Of PF-00345439 (Oxycodone) In Patients With Moderate To Severe Chronic Low Back Pain Or Osteoarthritis

DETAILED DESCRIPTION:
This study will evaluate: (a) the long-term safety of PTI-821 during a 12-month period; and (b) the long-term efficacy of PTI-821 by assessing pain intensity (PI), the quality of analgesia, and the global assessment of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are ≥ 18 and ≤ 75 years of age with moderate to severe pain in one or more hip or knee joint(s) caused by osteoarthritis for at least three months prior to the Baseline Visit or persistent moderate to severe low back pain for at least six months while regularly taking one or more of the following types of oral analgesic medication(s) prior to the Baseline Visit.
* Patient agrees to refrain from taking any opioid medications other than study drug during the study period. Patients must agree to report all non-opioid analgesic medications taken.
* Females who are postmenopausal, physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or IUD). If practicing an acceptable method of birth control, a negative urine pregnancy test result has been obtained at the Baseline Visit.

Exclusion Criteria:

* Patient has a positive urine drug screen at the Baseline Visit.
* Patient currently is on an opioid regimen with a daily opioid dose equivalent of oxycodone > 160 mg.
* Patient has major surgery planned during the proposed study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number and Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 12 months

SECONDARY OUTCOMES:
Percent change from baseline Pain Intensity Scale | baseline 1, 3, 6, 9 and 12 months
Quality of Analgesia - patient reported outcome of analgesia quality using ratings of excellent, very good, good, fair, or poor. | 1, 3, 6, 9 and 12 months
Global Assessment of Study Medication - patient reported outcome using ratings of excellent, very good, good, fair, or poor. | 1, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=PTI-821-CM&StudyName=Long-term%20safety%20of%20PF-00345439%20%28Oxycodone%29